CLINICAL TRIAL: NCT05400824
Title: Pathologies métaboliques et Infectieuses en Population générale à La Réunion : étude REUNION
Brief Title: Metabolic and Infectious Diseases in La Réunion (the REUNION Population-based Study)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C19-68; 2020A0209435 (Registry Identifier: IDRCB)
Record Dates: First submitted 2022-05-27; First posted 2022-06-02 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-05

CONDITIONS: Infectious Disease; Cardiovascular Diseases; General Population; Metabolic Disease
Keywords: epidemiology; risk factors; prevalence; cognitive impairment; dengue; hypertension; dyslipidemia; social inequalities; autonomous nervous system
MeSH Terms: conditions — Communicable Diseases; Cardiovascular Diseases; Metabolic Diseases; Cognitive Dysfunction; Dengue; Hypertension; Dyslipidemias | interventions — Blood Specimen Collection; DNA, B-Form; Defecation; Urination; Spirometry; Electrocardiography; Ultrasonography, Carotid Arteries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- general population: Observational study of 2000 adult men and women from the general population who will benefit from a free extensive health check up in La Reunion
  Interventions: Diagnostic Test: Blood, DNA, feces, urine, hair and skin microbiota collection

INTERVENTIONS:
Diagnostic Test: Blood, DNA, feces, urine, hair and skin microbiota collection — See above
  Other Names: Ewing test; Spirometry; EKG; cognitive, anxiety and depression tests; carotid ultrasound; pulse wave velocity measurement; ankle brachial index measurement

SUMMARY:
The aim of the present study is to determine the prevalence of cardiometabolic and infectious disease in La Reunion (french oversea department and region of France).

Known or suspected risk factor for these diseases will also be assessed, such as microbiota, cognitive impairement, social inequalities, and genetics.

DETAILED DESCRIPTION:
Overall, 2000 men and women will be recruited during two years for an extensive clinical examination including a microbiota, blood, hair and DNA collection, cognitive tests, autonomous nervous system assessment, spirometry, pulse wave velocity measurement, a carotid doppler echo tracking.

ELIGIBILITY:
Inclusion Criteria:

* 18-67 years
* given consent for genetic analysis,
* written consent for participating in the study

Exclusion Criteria:

* judicial protection or guardianship

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult men and women ramdomly selected from the voter registration lists in La Réunion island
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Prevalence of cardiometabolic diseases | cross sectional (at inclusion)
  Prevalence rates for diabetes, hypertension, obesity, dyslipidemia, smoking and subclinical atherosclerosis markers
Prevalence of infectious diseases | cross sectional (at inclusion)
  Seroprevalence rates for chikungunya, dengue, zika, covid19

CONTACTS AND LOCATIONS:
Overall Officials: Maxime COURNOT, MD, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France; Olivier MEILHAC, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France; Patrick MAVINGUI, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Centre Hospitalier Universitaire de La Réunion, La Réunion, Saint-Pierre, France

REFERENCES:
- See also: official website of the French National Institute for Health and Medical Research — http://www.inserm.fr